CLINICAL TRIAL: NCT02872168
Title: Identification of a New Metabolite of Furosemide in Humans
Acronym: PYPARK
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Philippe Le Corvoisier, professor, Henri Mondor University Hospital
Other Study IDs: 2014-A01789-38
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Treatment by Furosemide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not intervention — None. there is no modification in the treatment of patients. A urine collection is carry out in patients during the day of their enrolment.

SUMMARY:
Recent in-vitro and in-vivo studies performed by one of the investigators (ESO, ICMPE, UPEC, France) have recently allowed to synthetize a new and easy-to-synthesized chemical compound of the furosemide (pyridinium furosemide) during furosemide degradation by electro-Fenton or bioconversion. The biological properties of pyridinium furosemide are currently under investigation. Furosemide is a diuretics currently used in the treatment of patients with heart failure. The goal of the investigators is to assay pyridinium furosemide in urine of patients treated by furosemide to demonstrate that pyridinium is or not a metabolite of furosemide in humans. This study will contribute to assess the fate of pharmaceutical residues of furosemide in the environment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Written informed consent
3. Affiliation to social security
4. Known heart failure
5. Treatment by furosemide

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients treated by furosemide
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Assay of furosemide and pyridinium furosemide in urine of heart failure patients treated by furosemide | 1 day
  Assay of furosemide and pyridinium furosemide in urine of heart failure patients treated by furosemide

IPD SHARING:
Plan to Share IPD: No